CLINICAL TRIAL: NCT06915701
Title: "Evaluation of the Effect of Vitamin E (α-tocopherol) Supplementation on Clinical Activity and Inflammation in Patients With Rheumatoid Arthritis"
Brief Title: "Effect of Vitamin E (α-Tocopherol) on Clinical Activity and Inflammation in Rheumatoid Arthritis"
Acronym: VitE in RA
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Collaborators: Civil Hospital of Guadalajara (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI A-176/24
Record Dates: First submitted 2024-11-04; First posted 2025-04-08 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Antioxidant; Vitamin E
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Definition of patients: will be patients with RA deficient in vitamin E consumption (<15mg/day) , who are treated with conventional synthetic FARMEs (Methotrexate, Hydroxychloroquine, Leflunomide, Sulfasalazine and their combinations): The intervention group will take vitamin E 800mg/day, while the control group will take 200mg/day magnesium oxide placebo.
Who Masked: Participant, Investigator
Masking Description: Placebo use:
  Participants will be informed that they may be taking vitamin E or placebo. Both vitamin E and placebo will have similar excipients and be masked by similar packaging.
  - Double blind: It is important to minimize bias in the study that both the investigators involved as well as participants should be blinded as to who is receiving the active treatment and who is receiving the placebo. After the one-month period of supplementation and data collection, the study will be opened. An independent researcher to the project will be the one who keeps the information of the double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Treated with conventional synthetic FARMEs (Metrotexato, Hydroxychloroquine, Leflunomide, Sulfasalazina and their combinations) plus vitamin E 800mg/day.
  Interventions: Dietary Supplement: Will take vitamin E 800mg/day
- Control group (Placebo Comparator): Treated with conventional synthetic FARMEs (Metrotexato, Hydroxychloroquine, Leflunomide, Sulfasalazina and their combinations) plus the consumption of magnesium oxide 200mg/day in placebo form.
  Interventions: Drug: Will take 200mg/day magnesium oxide placebo.

INTERVENTIONS:
Dietary Supplement: Will take vitamin E 800mg/day — Patients with deficient vitamin E intake (<15mg/day), who are treated with conventional synthetic FARMEs (Metrotexato, Hydroxychloroquine, Leflunomide, Sulfasalazina and their combinations) plus vitamin E 800mg/day.
  Arms: Intervention group
Drug: Will take 200mg/day magnesium oxide placebo. — Patients with RA deficient in vitamin E intake (<15mg/day) , who are treated with conventional synthetic FARMEs (Metrotexato, Hydroxychloroquine, Leflunomide, Sulfasalazina and their combinations) plus the consumption of magnesium oxide 200mg/day in placebo form.
  Arms: Control group

SUMMARY:
The objective of this clinical trial is to determine whether α-tocopherol (vitamin E) supplementation decreases inflammation and clinical activity in patients with rheumatoid arthritis (RA).The main questions to be answered are:

* Is supplementation with vitamin E (α-tocopherol) for one month associated with decreased clinical activity and inflammation in patients with RA?

Researchers will compare α-tocopherol with a placebo (a look-alike substance containing no active ingredient) to see if α-tocopherol effectively reduces inflammation and clinical activity in patients with rheumatoid arthritis.

Participants will:

* Take two capsules (one in the morning and one in the afternoon) of either α-tocopherol or placebo every day for a month.
* Attend clinic visits at the start of the intervention (baseline) and at the end of the month for final check-ups and tests.
* Keep a diary to record your symptoms and how often you take α-tocopherol or placebo.

DETAILED DESCRIPTION:
Background:

Rheumatoid arthritis (RA) RA is one of the most common autoimmune diseases, characterized by chronic inflammation of the sinovia, mainly of the small joints of the hand, wrists and feet. Chronic inflammation can lead to the destruction of cartilage and joint bone, causing joint deformity, functional disability, depression and significant economic costs for the affected individual.

α-tocopherol acetate: The α-tocopherol acetate is the most widely used analogue in food supplements because of its esterification gives it stability. The main function is antioxidant preventing lipid oxidation of cell membranes for this reason α-tocopherol is considered a possible protector against diseases related to oxidative processes such as chronic diseasedegenerative diseases such as diabetes mellitus, cancer, cardiovascular disease, rheumatic disease, neurological disease and ageing.

Vitamin E in RA: The role of vitamin E as a therapy in combination with RA treatment has been studied in several studies. Studies in mouse models of laminarin-induced arthritis have shown that supplementation with α-tocopherol decreases the expression of pro-inflammatory cytokines such as IL-6, TNF-α and MMPs. However, the mechanisms involved are unknown. There are few studies in RA patients where the effect of supplementation with α-tocopherol has been analyzed. In clinical trials, it has been observed that from 3 weeks with supplementation of α-tocopherol decreases the scales of clinical activity in addition to morning stiffness and joint pain even biochemical parameters such as acute phase reactants such as pCr and ESR. However, the effect on pro-inflammatory cytokines, autoantibodies and antioxidant effect has not been analyzed.

Research question: Is supplementation with Vitamin E (α-tocopherol) for one month associated with decreased clinical activity and inflammation in patients with RA?

Specific objectives

1. Analyze the clinical characteristics and diet quality of RA patients
2. Determine serum autoantibody levels in RA patients
3. Quantify serum vitamin E levels before and after supplementation in both study groups (Vitamin E and placebo)
4. Compare clinical activity before and after supplementation in both study groups
5. Quantify serum concentration of pro-inflammatory cytokines IL1β, IL6 and TNF-α before and after supplementation in both study groups
6. Determine antioxidant capacity before and after supplementation in both study groups
7. Associate vitamin E levels with clinical and inflammatory parameters of patients with RA

Hypothesis :

There is an association between supplementation with vitamin E (α-tocopherol) and decreased clinical activity and inflammation in patients with RA from western Mexico

Methodological design:

a) Study type - Clinical, randomized, controlled and double-blind trial.

Research sites:

* Institute of Biomedical Sciences (IICB) of the University Center for Health Sciences (CUCS)
* Laboratory for Clinical Analysis and Translational Research (LACIT), at the University Center for Exact Sciences and Engineering (CUCEI)
* Rheumatology Service of the Civil Hospital "Fray Antonio Alcalde" in Guadalajara, Jalisco.

Time to develop: January 2025 to January 2027.

Sample size:

The statistical formula of two averages was used for the calculation of the sample size. The calculations were made with data from the corresponding 2001 clinical trial of Mona Helmy and colleagues, resulting in a sample size of 19 patients plus an increase of 20% to cover possible losses. Having 23 patients for control and intervention group. Both groups with RA of the Rheumatology Service of the Civil Hospital "Fray Antonio Alcalde" in Guadalajara, Jalisco.

Variables Independent variables

* Vitamin E Dependent variables
* Inflammatory cytokines (IL-1β, IL-6 and TNF-α). Antioxidant capacity:( DPPH, ABTS, FRAP and ORAC). Clinical evolution: DAS-28. Acute phase reactants: pCr and ESR. Auto-antibodies: Anti-ccp and rheumatoid factor.

Biosafety considerations:

This study will apply the guidelines set out in the Mexican Official Standards, NOM-052-SEMARNAT-2005, NOM-054-SEMARNAT-1993 and NOM-087-ECOL-SSA1-2002 that refer to classification, Handling, storage and disposal of hazardous waste, chemical reagents and biological-infectious wastes, in order to ensure the protection of people in contact with them and the environment.

Ethical considerations:

The project will be carried out in accordance with the ethical standards and principles for medical research on human beings, as set out in the Declaration of Helsinki, which were last reviewed at the 64th General Assembly, Fortaleza, Brazil, October 2013, which refers to ethical principles for medical research in humans.

ELIGIBILITY:
Inclusion criteria:

* Female sex
* RA classification (ACR/EULAR 2010)
* Early RA 2 years
* Treatment with conventional synthetic FARMEs (Metrotexato, Hydroxychloroquine, Leflunomide, Sulfasalazina and their combinations)
* DAS28 ≥3.2
* Vitamin E intake deficiency (<15mg/day)
* No comorbidities
* Age > 18 years
* Voluntary participation and informed consent.

Exclusion Criteria:

* Liver and kidney disease
* Overlap syndrome
* Coagulation disorders
* Pregnancy
* Consumption of supplements (iron, vitamin E, and K), and medications such as acetylsalicylic acid, amlodipine, estrogen, glucocorticoids and drugs used to treat dyslipidemias in the last three months.

Elimination Criteria:

* Errors in administration of the 20% supplement
* Adverse effects of the supplement
* Pregnancy during the study
* Insufficient blood sample
* Voluntary withdrawal of informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 46 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Levels of vitamin E | Exchange measures: Baseline and 1 month.
  Adequacy:12 and 20 µg/mL (27.9-46.4 µmol/L). Insufficiency: 5 and 12 µg/mL (11.6-27.9 µmol/L). Minor deficiency of: 5 µg/mL (11.6 µmol/L).

SECONDARY OUTCOMES:
Twenty-four hour reminder "questionnaire" (Recommended Daily Intake of Vitamin E) | Exchange measures: Baseline and 1 month.
  Twenty-four hour reminder:
  Will be done by the nutritionist, who will ask about the food consumed on the previous day to evaluate the quality of the diet and vitamin E consumption. The twenty-four hour reminder is a subjective method, retrospective, conducted through a face-to-face or telephone interview. This method is based on accurately remembering, describing and quantifying the food consumed one day before the consultation. All the patient's dietary intake throughout the day should be described in detail.
  > 19 years old. 15 mg daily.
Levels of: Proinflammatory cytokines ( IL-1β , IL-6 and TNF-α ) | Exchange measures: Baseline and 1 month.
  Units: pg/ml
Antioxidant capacity: (DPPH, ABTS, FRAP and ORAC) | Exchange measures: Baseline and 1 month.
  Units: μmol EQ trolox/μL sample
Index DAS-28 | Exchange measures: Baseline and 1 month.
  Remission: < 2.6 Low activity: 2.6 <3.2 Moderate: 3.2 < 5.1 High: 5.1
C-reactive protein (pCr) | Exchange measures: Baseline and 1 month.
  19-49 years < 3.33 mg/L 50-64 years < 8.50 mg/L
Erythrocyte sedimentation rate (ESR) | Exchange measures: Baseline and 1 month.
  20 mm/hr
Auto- antibodies: Anti-CCP | Exchange measures: Baseline and 1 month.
  Positive: > 5 U/mL Positive highs > 3 times cut-off value
Rheumatoid factor | Exchange measures: Baseline and 1 month.
  Positive > 20 IU/mL Positive highs > 3 times the cut-off value

CONTACTS AND LOCATIONS:
Overall Officials: Christian Johana J Baños Hernández, D.Sc., Principal Investigator — University of Guadalajara
Locations (2):
- Mexico (2):
  - Civil Hospital of Guadalajara, Guadalajara, Jalisco
  - Universidad de Guadalajara, Guadalajara, Jalisco

IPD SHARING:
Plan to Share IPD: No
No: There is no plan to make IPD available.

REFERENCES:
- [Background] Kim KW, Kim BM, Won JY, Min HK, Lee SJ, Lee SH, Kim HR. Tocotrienol regulates osteoclastogenesis in rheumatoid arthritis. Korean J Intern Med. 2021 Mar;36(Suppl 1):S273-S282. doi: 10.3904/kjim.2019.372. Epub 2020 Jun 19. PMID 32550719
- [Background] Hama S, Kirimura N, Obara A, Takatsu H, Kogure K. Tocopheryl Phosphate Inhibits Rheumatoid Arthritis-Related Gene Expression In Vitro and Ameliorates Arthritic Symptoms in Mice. Molecules. 2022 Feb 20;27(4):1425. doi: 10.3390/molecules27041425. PMID 35209214
- [Background] Al-Okbi SY. Nutraceuticals of anti-inflammatory activity as complementary therapy for rheumatoid arthritis. Toxicol Ind Health. 2014 Sep;30(8):738-49. doi: 10.1177/0748233712462468. Epub 2012 Oct 26. PMID 23104728
- [Background] Zhang T, Yi X, Li J, Zheng X, Xu H, Liao D, Ai J. Vitamin E intake and multiple health outcomes: an umbrella review. Front Public Health. 2023 Jul 13;11:1035674. doi: 10.3389/fpubh.2023.1035674. eCollection 2023. PMID 37522003
- [Background] Glowka AK, Kowalowka M, Burchardt P, Komosa A, Kruszyna L, Andrusiewicz M, Przyslawski J, Karazniewicz-Lada M. Selected Psychosocial Factors, Nutritional Behavior, and the Analysis of Concentrations of Selected Vitamins in Patients with Cardiovascular Diseases. Nutrients. 2024 Jun 14;16(12):1866. doi: 10.3390/nu16121866. PMID 38931221
- [Background] Galli F, Azzi A, Birringer M, Cook-Mills JM, Eggersdorfer M, Frank J, Cruciani G, Lorkowski S, Ozer NK. Vitamin E: Emerging aspects and new directions. Free Radic Biol Med. 2017 Jan;102:16-36. doi: 10.1016/j.freeradbiomed.2016.09.017. Epub 2016 Nov 2. PMID 27816611
- [Background] Lewis ED, Meydani SN, Wu D. Regulatory role of vitamin E in the immune system and inflammation. IUBMB Life. 2019 Apr;71(4):487-494. doi: 10.1002/iub.1976. Epub 2018 Nov 30. PMID 30501009
- [Background] Kemnic TR, Coleman M. Vitamin E Deficiency. 2023 Jul 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519051/ PMID 30085593
- [Background] Brigelius-Flohe R. Vitamin E research: Past, now and future. Free Radic Biol Med. 2021 Dec;177:381-390. doi: 10.1016/j.freeradbiomed.2021.10.029. Epub 2021 Oct 29. PMID 34756995
- [Background] Mohd Zaffarin AS, Ng SF, Ng MH, Hassan H, Alias E. Pharmacology and Pharmacokinetics of Vitamin E: Nanoformulations to Enhance Bioavailability. Int J Nanomedicine. 2020 Dec 8;15:9961-9974. doi: 10.2147/IJN.S276355. eCollection 2020. PMID 33324057
- [Background] Traber MG, Head B. Vitamin E: How much is enough, too much and why! Free Radic Biol Med. 2021 Dec;177:212-225. doi: 10.1016/j.freeradbiomed.2021.10.028. Epub 2021 Oct 23. PMID 34699937
- [Background] Mueller AL, Payandeh Z, Mohammadkhani N, Mubarak SMH, Zakeri A, Alagheband Bahrami A, Brockmueller A, Shakibaei M. Recent Advances in Understanding the Pathogenesis of Rheumatoid Arthritis: New Treatment Strategies. Cells. 2021 Nov 4;10(11):3017. doi: 10.3390/cells10113017. PMID 34831240
- [Background] Orellana C, Saevarsdottir S, Klareskog L, Karlson EW, Alfredsson L, Bengtsson C. Oral contraceptives, breastfeeding and the risk of developing rheumatoid arthritis: results from the Swedish EIRA study. Ann Rheum Dis. 2017 Nov;76(11):1845-1852. doi: 10.1136/annrheumdis-2017-211620. Epub 2017 Aug 17. PMID 28818831
- [Background] Padyukov L. Genetics of rheumatoid arthritis. Semin Immunopathol. 2022 Jan;44(1):47-62. doi: 10.1007/s00281-022-00912-0. Epub 2022 Jan 27. PMID 35088123
- [Background] Busch R, Kollnberger S, Mellins ED. HLA associations in inflammatory arthritis: emerging mechanisms and clinical implications. Nat Rev Rheumatol. 2019 Jun;15(6):364-381. doi: 10.1038/s41584-019-0219-5. PMID 31092910
- [Background] Munoz-Valle JF, Padilla-Gutierrez JR, Hernandez-Bello J, Ruiz-Noa Y, Valle Y, Palafox-Sanchez CA, Parra-Rojas I, Gutierrez-Urena SR, Rangel-Villalobos H. PTPN22 -1123G>C polymorphism and anti-cyclic citrullinated protein antibodies in rheumatoid arthritis. Med Clin (Barc). 2017 Aug 10;149(3):95-100. doi: 10.1016/j.medcli.2017.01.025. Epub 2017 Mar 11. English, Spanish. PMID 28291534
- [Background] Almutairi K, Nossent J, Preen D, Keen H, Inderjeeth C. The global prevalence of rheumatoid arthritis: a meta-analysis based on a systematic review. Rheumatol Int. 2021 May;41(5):863-877. doi: 10.1007/s00296-020-04731-0. Epub 2020 Nov 11. PMID 33175207
- [Background] Moreno-Montoya J, Alvarez-Nemegyei J, Sanin LH, Perez-Barbosa L, Trejo-Valdivia B, Santana N, Goycochea-Robles MV, Cardiel MH, Riega-Torres J, Maradiaga M, Burgos-Vargas R, Pelaez-Ballestas I; GEEMA (Grupo de Estudio Epidemiologico de Enfermedades Musculo Articulares). Association of regional and cultural factors with the prevalence of rheumatoid arthritis in the Mexican population: a multilevel analysis. J Clin Rheumatol. 2015 Mar;21(2):57-62. doi: 10.1097/RHU.0000000000000223. PMID 25710855
- [Background] Castillo-Canon JC, Trujillo-Caceres SJ, Bautista-Molano W, Valbuena-Garcia AM, Fernandez-Avila DG, Acuna-Merchan L. Rheumatoid arthritis in Colombia: a clinical profile and prevalence from a national registry. Clin Rheumatol. 2021 Sep;40(9):3565-3573. doi: 10.1007/s10067-021-05710-x. Epub 2021 Mar 27. PMID 33772350
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Cush JJ. Rheumatoid Arthritis: Early Diagnosis and Treatment. Med Clin North Am. 2021 Mar;105(2):355-365. doi: 10.1016/j.mcna.2020.10.006. PMID 33589108

DOCUMENTS (1):
  • Study Protocol (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT06915701/Prot_000.pdf